CLINICAL TRIAL: NCT00001928
Title: Intravenous Levodopa in Parkinsonism
Brief Title: Intravenous Levodopa for the Diagnosis of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990072; 99-N-0072
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-03

CONDITIONS: Parkinson Disease
Keywords: Diagnosis; Infusion; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Disease; Parkinsonian Disorders

SUMMARY:
Patients with Parkinson's disease have low levels of the neurotransmitter dopamine. Dopamine is responsible for motor function and normal physical activity. Patients with Parkinson's disease typically suffer from tremors, rigid muscles, stooped postures, and walk with a shuffle. The drug levodopa acts as a replacement for dopamine and has been has been used effectively for over 30 years as treatment for Parkinsons disease. Because of its effectiveness, levodopa has been used to distinguish Parkinson's disease from other conditions that may resemble Parkinson's disease.

Traditionally, levodopa has been given as a pill. In this study, researchers would like to inject levodopa directly into a vein (intravenous) in order to diagnose cases of Parkinson's disease. This method provides immediate results and allows doctors to adjust the dose of levodopa very carefully. Because the intravenous method of giving levodopa is less practical than oral medication, it is not an available alternative for the routine treatment of Parkinson's disease. However, it may be useful for faster diagnosis of the disease and for determining effective doses of oral medication.

DETAILED DESCRIPTION:
A positive response to levodopa is now considered a condition sine qua non for the diagnosis of idiopathic Parkinson's disease. Under this protocol, patients with parkinsonism of uncertain etiology will be tested for their motor response to intravenous levodopa to aid in the diagnosis of Parkinson's disease. This protocol regulates and stipulates the acute administration of intravenous levodopa and associated safety issues.

ELIGIBILITY:
All patients will have parkinsonism of undetermined etiology.

Males and females between the ages of 18 and 85 are eligible for the study.

No presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risks, specifically those who have the following: a history of convulsive, hepatic, or renal disorders; currently receiving treatment for myocardial infarction, arrhythmia or cardiac failure; and pregnant women or anyone not practicing an effective means of birth control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1999-03; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fabbrini G, Juncos J, Mouradian MM, Serrati C, Chase TN. Levodopa pharmacokinetic mechanisms and motor fluctuations in Parkinson's disease. Ann Neurol. 1987 Apr;21(4):370-6. doi: 10.1002/ana.410210409. PMID 3579222
- [Background] Mouradian MM, Juncos JL, Fabbrini G, Chase TN. Motor fluctuations in Parkinson's disease: pathogenetic and therapeutic studies. Ann Neurol. 1987 Oct;22(4):475-9. doi: 10.1002/ana.410220406. PMID 3435068
- [Background] Fabbrini G, Mouradian MM, Juncos JL, Schlegel J, Mohr E, Chase TN. Motor fluctuations in Parkinson's disease: central pathophysiological mechanisms, Part I. Ann Neurol. 1988 Sep;24(3):366-71. doi: 10.1002/ana.410240303. PMID 3228270